CLINICAL TRIAL: NCT02415010
Title: A Post-Market Clinical Follow-Up Study to Confirm Clinical Performance and Safety of the Codman Enterprise® 2 Vascular Reconstruction Device in the Endovascular Treatment of Intracranial Aneurysms
Brief Title: Post-Market Clinical Follow-Up Study to Confirm Clinical Performance and Safety of the Codman Enterprise® 2 Vascular Reconstruction Device in the Endovascular Treatment of Intracranial Aneurysms
Acronym: SUNRISE-2
Status: Terminated | Type: Observational
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NV-PMK-1401
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Enterprise 2 Vascular Reconstruction Device — Stenting Assisted coiling procedure

SUMMARY:
The objective of this Post-Market Clinical Follow-up (PMCF) is to confirm the performance and safety of the Codman Enterprise® 2 when used in conjunction with endovascular coil embolization of ruptured or non-ruptured intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years old.
2. Subjects with non-ruptured or ruptured intracranial aneurysm that is referred for endovascular treatment.
3. Parent vessel with a diameter of ≥ 2.0 mm and ≤ 4 mm.
4. Subject understands the nature of the procedure and provides voluntary written informed consent in accordance with the requirements of this study protocol.
5. Subject is willing to participate in the telephone follow-ups and to return to the investigational site for the post-procedure follow-up evaluations.

Exclusion Criteria:

1. Angiogram demonstrating that the aneurysm is not appropriate for endovascular treatment (i.e.: severe intracranial vessel tortuosity, stenosis, intracranial vasospasm not responsive to medical therapy).
2. Mycotic or traumatic aneurysm.
3. Arteriovenous malformation (AVM) in the territory of the target aneurysm.
4. Two or more aneurysms (>2mm) in associated distribution.
5. Hunt and Hess Scale (HHS) of IV or V at inclusion for subject with ruptured aneurysms.
6. Life expectancy of less than 6 months as determined by the treating physician.
7. A planned staged procedure (i.e. a procedure where entire treatment with the devices (e.g. coils/stents) is completed over separate sessions).
8. Previous neuro-interventional or neuro-surgical procedure of any kind within 30 days prior to the study procedure.
9. Intracranial mass (tumor, abscess, or other infection), or undergoing radiation therapy for carcinoma or sarcoma of the head or neck region.
10. Unsuitable for the antithrombotic and/or anticoagulant therapies
11. Serum creatinine level > 2.5 mg/dl within 7 days prior to index procedure
12. Known hypersensitivity or allergies to cobalt, nitinol metal, nickel, or sensitivity to contrast media,
13. Evidence of an acute myocardial infarction (MI) within 30 days prior to the index procedure.
14. Uncontrolled atrial fibrillation or known cardiac disorders likely to be associated with cardioembolic symptoms.
15. Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with both ruptured and non-ruptured aneurysms will be enrolled into the study, with a parent vessel diameter of ≥ 2.0 mm and ≤ 4 mm
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Major Ipsilateral Stroke and/or Death due to related neurological event in subjects with a non-ruptured aneurysm. | 6 months
  any a new neurological event, which is ipsilateral and in the vascular distribution territory of the stenting procedure and that results in an increase of ≥ 4 on the National Institute of Health Stroke Scale (NIHSS), as compared to baseline and persists for greater than 24 hours

SECONDARY OUTCOMES:
Incidence of Successful Aneurysm treatment without retreatment | 6 Months
  aneurysms categorized as adequate occlusion (i.e., scored as complete [100%] or near completely occluded [90-99%]), without additional procedures for treatment of the aneurysm since the index procedure.
Incidence of Successful Aneurysm treatment | 12 months
  aneurysms categorized as adequate occlusion (i.e., scored as complete [100%] or near completely occluded [90-99%]), without additional procedures for treatment of the aneurysm since the index procedure.
Incidence of Aneurysm Recanalization | 6 & 12 Months
  any increase in aneurysm filling, compared to the previous study-specified angiographic assessment, resulting in a change in (i.e., worsening of) the 3-point scale.
Incidence of Retreatment | 6 & 12 Months
  aneurysms with any additional treatment of the target aneurysm after the index procedure (regardless of whether retreatment is by surgery or endovascular treatment) due to recanalization, rupture, bleeding or staged procedure.
Incidence of New Neurological Deficits | 30 Days, 6 & 12 Months
  subjects who have an increase in mRS greater than 2 from baseline related to stroke or death
Incidence of Major Ipsilateral Stroke and/or Death due to related neurological event | 30 Days and 12 Months
  any a new neurological event, which is ipsilateral and in the vascular distribution territory of the stenting procedure and that results in an increase of ≥ 4 on the National Institute of Health Stroke Scale (NIHSS), as compared to baseline and persists for greater than 24 hours
Incidence of Parent Vessel Thrombosis | 6 & 12 Months
  parent vessel arteries in which thrombosis was documented by an angiogram
Incidence of Parent Vessel Stenosis | 6 & 12 Months
  parent vessel arteries in which stenosis was documented by an angiogram,
Incidence of Stent Movement/Migration | 6 & 12 Months
  parent artery in which CODMAN Enterprise® 2 migration was documented from the index procedure until completion of the follow-up visit.
Frequency of Adverse Events | 6 & 12 Months
  Occurence of any AE related to device/procedure/disease

CONTACTS AND LOCATIONS:
Overall Officials: J FIEHLER, MD-PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (10):
- Germany (5):
  - Helios Klinikum Berlin, Berlin
  - Universitätslklinikum der Ruhr Universität Bochum, Bochum
  - Universitätsklinikum Hamburg Eppendorf, Eppendorf
  - Asklepios Klinik Atona, Hamburg
  - Universitätsklinikum Schl.-Holst. Campus Lübeck, Lübeck
- Hospital Universitario de Navarra, Pamplona, Spain
- Switzerland (2):
  - Inselspital-Universitätsspital Bern, Bern
  - Hôpitaux Universitaires de Genève, Geneva
- United Kingdom (2):
  - Spire Leeds Hospital, Leeds
  - Queen's Hospital of Romford, Romford